CLINICAL TRIAL: NCT00332150
Title: Mothers' Approach to Clinical Research Amongst Their Preterm or Healthy Newborns
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ayala Maayan, Sehba Medical Center
Other Study IDs: SHEBA-06-4076-AM-CTIL
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Parents Approval to Research
Keywords: parents; newborn; clinical trials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Parental approval to enroll their sick children in clinical research was studied. However, the motivation of parents to enroll healthy children and/or babies was not yet studied. The importance of clinical research among the healthy population is of extreme value. The aim of this study is to assess the motivation, medical trust and other factors influencing parents' decision to enroll their healthy baby in a clinical study.

DETAILED DESCRIPTION:
Mothers to either healthy full-term babies post delivery or preterms will be asked to anonymously answer a questionnaire. The questionnaire includes demographic data, questions regarding their approach to medical issues, factors that influence her to enroll her baby in a research trial (different research types, different benefits from the research and fears). Finally, the mother will be asked if she will be willing to enroll her baby to on-going studies in the department.

ELIGIBILITY:
Inclusion Criteria:

* Mothers to healthy newborns during hospital stay after delivery, and mothers of preterm infants during their hospitalization in NICU.

Exclusion Criteria:

* Mothers of sick newborns (respiratory distress, receiving IV infusion, etc.) who are in the special care for newborns.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2006-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Maayan, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Zupancic JA, Gillie P, Streiner DL, Watts JL, Schmidt B. Determinants of parental authorization for involvement of newborn infants in clinical trials. Pediatrics. 1997 Jan;99(1):E6. doi: 10.1542/peds.99.1.e6. PMID 9096174
- [Derived] Maayan-Metzger A, Kedem-Friedrich P, Kuint J. Motivations of mothers to enroll their newborn infants in general clinical research on well-infant care and development. Pediatrics. 2008 Mar;121(3):e590-6. doi: 10.1542/peds.2007-1571. PMID 18310179